CLINICAL TRIAL: NCT02430493
Title: A Multi-Centre, Prospective Cohort, Non-Interventional Study About Evaluation on the Safety of Ticagrelor Among Chinese ACS Patients
Brief Title: Evaluation on the Safety of Ticagrelor Among Chinese ACS Patients
Acronym: YingLong
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130R00026
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: ACS
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ticagrelor: Chinese subjects aged over 18, diagnosed as ACS and treated with ticagrelor at least one tablet

SUMMARY:
The primary objective is to describe the safety and tolerability of ticagrelor, by assessment of adverse events (characteristics, reporting rate, severity, relationship and risk factors), especially the bleeding events as defined in 8.1 and other serious adverse events (SAEs) during 1-year follow up in Chinese acute coronary syndrome (ACS) patients.

DETAILED DESCRIPTION:
The trial is a multi-centre, prospective cohort, non-interventional study to be conducted in the department of cardiology from approximately 20 tier-2 or 3 hospitals, China. The study requires Chinese subjects aged over 18, diagnosed as ACS and treated with ticagrelor at least one tablet from the department of cardiology in the around 20 tier-2 or 3 hospitals. The subjects will be tracked up to 1 month after the discontinuation of ticagrelor for AE events and 1 year after enrollment for major cardiovascular events. This is an observational study. The prescribing doctor is in charge of prescribing or discontinuation ticagrelor. The investigator in an observational study may not intervene in the treatment. All 1000 subjects' related data will be collected

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of informed consent prior to any study specific procedures 2. Chinese female or male aged at least 18 years 3. Index event of non-ST or ST segment elevation ACS. 4. Taken with ticagrelor at least one tablet before enrollment.

Exclusion Criteria:

-1. Participation in another clinical study with an investigational product during the last 6 months.

2. Previous enrolment in the present study; 3. Allergy or any other contraindication to ticagrelor as described in ticagrelor China PI.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese subjects aged over 18, diagnosed as ACS and treated with ticagrelor at least one tablet from the department of cardiology in the around 20 tier-2 or 3 hospitals.
Sampling Method: Probability Sample
Enrollment: 1066 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ticagrelor, by assessment of adverse events, especially the bleeding events and other SAEs during 1-year follow up in Chinese ACS patients. | 1 year
  a) Incidence of post-authorization adverse events including characteristics, reporting rate, severity, relationship and risk factors among Chinese ACS patients with ticagrelor during 1-year follow up b) PLATO-defined fatal/life-threatening bleedings during 1-year follow up in Chinese ACS patients treated with ticagrelor. c) PLATO-defined major bleedings during 1-year follow up in Chinese ACS patients treated with ticagrelor. d) PLATO-defined major + minor bleedings during 1-year follow up in Chinese ACS patients treated with ticagrelor. e) PLATO-defined major + minor + minimal bleedings during 1-year follow up in Chinese ACS patients treated with ticagrelor. f) Serious adverse events other than bleeding during 1-year follow up in Chinese ACS patients treated with ticagrelor

SECONDARY OUTCOMES:
Incidence of major cardiovascular (CV) events during 1-year follow up in Chinese ACS patients treated with ticagrelor. | 1 year
  Major CV events including CV death, MI and Stroke, during 1 year follow up in Chinese ACS patients treated with ticagrelor. Incidence of post-authorization adverse events among specific patients groups from Chinese ACS patients with ticagrelor. Survival free of major CV events among Chinese ACS patients with ticagrelor. Proportion of patients with discontinuation or interruption of ticagrelor and the reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Principal Investigator — Beijing Anzhen Hospital
Locations (15):
- China (15):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Huai'an
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Suqian
  - Research Site, Tai’an
  - Research Site, Wuhan
  - Research Site, Xuzhou
  - Research Site, Zhengzhou

REFERENCES:
- [Background] Li J, Li X, Wang Q, Hu S, Wang Y, Masoudi FA, Spertus JA, Krumholz HM, Jiang L; China PEACE Collaborative Group. ST-segment elevation myocardial infarction in China from 2001 to 2011 (the China PEACE-Retrospective Acute Myocardial Infarction Study): a retrospective analysis of hospital data. Lancet. 2015 Jan 31;385(9966):441-51. doi: 10.1016/S0140-6736(14)60921-1. Epub 2014 Jun 23. PMID 24969506
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Derived] Du X, Zheng Y, Yang P, Ma S, Yu Z, Su X, Ge J, Leonsson-Zachrisson M, Wang X, Sun J, Bai L, Ma CS; YINGLONG study investigators. YINGLONG: A Multicenter, Prospective, Non-Interventional Study Evaluating the Safety and Tolerability of Ticagrelor in Chinese Patients with Acute Coronary Syndrome. Adv Ther. 2019 Jul;36(7):1595-1605. doi: 10.1007/s12325-019-00972-z. Epub 2019 May 22. PMID 31119693
- See also: D5130R00026 synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3711&filename=D5130R00026synopsis.pdf